CLINICAL TRIAL: NCT02954926
Title: Effect of Intravenous Immunoglobulin in Prevention of Preterm Neonatal Sepsis
Brief Title: Intravenous Immunoglobulin in Prevention of Preterm Neonatal Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Mahboobi, Resident of internal medicine, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUMS.REC.1394.162
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVIG (Experimental): IVIG at a dose of 500mg/kg within 12 h and 3 days of birth
  Interventions: Drug: IVIG
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: IVIG — IVIG at a dose of 500mg/kg within 12 h and 3 days of birth
  Arms: IVIG

SUMMARY:
Majority of healthcare authorities believe that due to the methodological weakness and small number of patients in conducted therapeutic trials, the evidences are insufficient to support the efficacy of intravenous immunoglobulin (IVIG) in prevention of preterm neonatal sepsis. The objective of this research is to determine the effect of intravenous immunoglobulin in prevention of preterm neonatal sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Born alive before 37 weeks of pregnancy (preterm neonates)
* Under 2500 g at birth

Exclusion Criteria:

* lethal anomaly
* congenital heart disease
* TORCH infection
* severe asphyxia

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Mortality | 7 days
  Death from sepsis or its related complications

SECONDARY OUTCOMES:
Total number of days of hospitalization | 7 days
  Duration of hospitalization
Intraventricular Hemorrhage | 7 days
  occurrence of Intraventricular Hemorrhage
Necrotizing enterocolitis | 7 days
  occurrence of Necrotizing enterocolitis
Bronchopulmonary dysplasia | 7 days
  occurrence of Bronchopulmonary dysplasia

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Mohammadi hospital, Bandar Abbas, Hormozgan, Iran

IPD SHARING:
Plan to Share IPD: No